CLINICAL TRIAL: NCT02504060
Title: Multicenter Randomized Double-blind Placebo-controlled Clinical Trials to Evaluate the Clinical Efficacy and Safety of N-acetyl Glucosamine Capsule for Irritable Bowel Syndrome With Diarrhea (IBS-D) Treatment
Brief Title: Clinical Trials of N-acetyl Glucosamine Capsule for IBS-D Treatment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Liujunkang, The director of microecological pharmaceutical research, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMMUBC; dongying (Other Grant/Funding Number: Dongying leader pharmaceutical co.,LTD)
Record Dates: First submitted 2015-07-16; First posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: diarrhea; abdominal pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea; Abdominal Pain | interventions — Acetylglucosamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Starch capsule (Placebo Comparator): During the 12- weeks treatment phase of the study, the daily dose of 3 tablets will be taken 30 minutes after breakfast, lunch and supper.
  Interventions: Drug: Starch Placebo
- N-acetyl-D-glucosamine (Experimental): During the 12- weeks treatment phase of the study, the daily dose of 100mg*3 (3 tablets) will be taken 30 minutes after breakfast, lunch and supper.
  Interventions: Drug: N-acetyl-D-glucosamine

INTERVENTIONS:
Drug: Starch Placebo
  Arms: Starch capsule
Drug: N-acetyl-D-glucosamine
  Other Names: Atysamine(ATSM)
  Arms: N-acetyl-D-glucosamine

SUMMARY:
This study is a randomized double-blind placebo-controlled clinical trail to evaluate the clinical efficacy and safety of 1.1 chemical drugs N-acetyl-D-glucosamine on Chinese IBS-D patients coming from thirty- six centers in Chinese. 720 IBS-D patients (360 for treatment group, 360 for placebo group) in this research are accord with the Rome III diagnostic criteria, screening/import period pain intensity scores of the NRS(numerical rating scale) week mean value are 3.0 plus and the days which at least more than one time a stool type are 6 or 7 type over 2 days/week. Test cycle includes screening/import period (2 weeks), open treatment period (12 weeks), follow-up period (2 weeks). The main outcome measures are pain intensity (NRS score 11 point scale) and stool type ( Bristol type), and secondary endpoints included overall symptoms sensory scores, defecation frequency, abdominal distension, defecation urgency and quality of life parameters (IBS-QOL scale).

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed the informed consent form.
* Man or woman, aged 18 to 65 years, inclusive.
* Based on the Roman III diagnostic criteria for diagnosis of IBS-D subjects, recurrent abdominal pain accompanied with abdominal discomfort or not, monthly attack within the past 3months at least 3 days. With two or more of the following three kinds of symptoms:

At least a portion of the time abdominal pain or defecate increase when discomfort.

At least a portion of the time abdominal pain or the row of loose stools when discomfort.

At least a portion of the time abdominal pain or discomfort improved after defecation.

Symptoms for at least 6 months before diagnosis.

* Screening/import period pain intensity scores of the NRS week mean value are 3.0 plus and the days which at least more than one time a stool type are 6 or 7 type over 2 days per week.
* During the screening period，patients should answer the questions of electronic log completely following the requirements for 10days or more.
* Patients are willing to stop drugs for abdominal symptoms or diarrhea which are in violation of the scheme, and take medicine prescribed in the scheme.
* Patients agree to not change the lifestyle significantly that may affect the symptoms of IBS-D from signing up the Informed Consent Form to the last experiment.
* The illness recured after a normal colonoscopy report within one year that was provided by this hospital or a grade first class teaching hospital, include polyp of colon (less than 3mm,the number of less than 5) patients who taked therapeutic endoscopy and recurrenced within one year; or those that get a normal colonoscopy report in this hospital or a grade first class teaching hospital before screening but have a history of bowel preparation, should be chosen when next attack.

Exclusion Criteria:

* History of organic gastrointestinal diseases: Chronic pancreatitis (cp), inflammatory bowel disease, intestinal tuberculosis, malabsorption syndrome, celiac disease, gastrointestinal tumor, or other organic diseases etc.
* History of abdominal and pelvic surgery ( not including appendectomy and intestinal polyposis (<3mm) after treatment within one year ).
* The non-intestinal disease of digestive system such as Peptic ulcer, tuberculous peritonitis, cirrhosis etc.
* Heart, lung, kidney and other important organs have severe lesions, immune regulatory disease, metabolic disease (diabetes, thyroid disease) or malignant tumor, reproductive system diseases such as ovarian cysts, endometriosis, etc.
* Laboratory tests or Electrocardiogram were significantly abnormal, and judging by the researchers may damage the patient safety or successful completion of the clinical research:

Male hemoglobin <120g/L, female hemoglobin <100g/L;

Male serum creatinine≥133umol/L, female serum creatinine≥124umol/L; or creatinine clearance rate≤60ml/min;

Chronic liver disease and/or abnormal liver function, defined as AST (aspartate aminotransferase) > 1.5 x ULN (Upper Limit Of Normal) and/or ALT (alanine aminotransferase) > 1.5 x ULN and/or total bilirubin > 1.5x ULN;

* Serious psychiatric patients( Hamilton Depression Scale scores>20).
* History of drug abuse or alcohol abuse.
* Allergic to this study drug.
* Concomitant medication is unable to stop or use continuously for more than a week but affect the gastrointestinal movement and function in the experiment, such as antibiotic drugs, the drugs of regulating the intestinal microecology, parasympathetic inhibitors, muscle relaxants, antidiarrheal, opiates, etc.
* Do not fill in the electronic log of one week before entering the group (-1 week) completely.
* Pregnant or lactating women
* Is participating in clinical trials or have finished it less than 3 months.
* Other researchers think not suitable for the list.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Abdominal Pain Intensity | one and a half years
  As measured by numerical rating scale
Stool Consistency | one and a half years
  As measured by Bristol ' s scale

SECONDARY OUTCOMES:
General symptoms feel grading | one and a half years
  As measure by patient reported outcome measures
defecation frequency | one and a half years
  As measure by patient reported outcome measures
abdominal distension | one and a half years
  As measure by patient reported outcome measures
Defecation urgency | one and a half years
  As measure by patient reported outcome measures
life quality parameters | one and a half years
  As measure by healthy survey, SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Junkang Liu, Doctor, Study Chair — Third MMU
Locations (1):
- Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China